CLINICAL TRIAL: NCT03939494
Title: Enhancing Effectiveness Of Existing Weight Management Programs For Teens With Severe Obesity: A 6-Month Feasibility Pilot
Brief Title: Healthy Weight for Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Helen DeVos Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-4028
Record Dates: First submitted 2019-04-11; First posted 2019-05-06 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Intervention (Experimental): This arm receives 26 hours of telehealth encounters with a registered dietitian in conjunction with their normal clinic/program care.
  Interventions: Behavioral: Telehealth Encounter
- Standard of Care Control (No Intervention): This arm will participate in their normal clinic/program routine.

INTERVENTIONS:
Behavioral: Telehealth Encounter — Contact will be made with participants via Face Time or Skype.
  Arms: Telehealth Intervention

SUMMARY:
POWER is uniquely positioned to evaluate characteristics of multi-component PWM programs that are associated with "favorable" health outcomes for treatment-seeking youth with obesity. The POWER Data Coordinating Center developed ranking reports of the 33 participating sites based on weight status change at 6 months. An in-depth review of program design of 4 "top-performing" sites was conducted. A unique feature identified was offering an individual program orientation session to patient-families prior to the start of the multi-component PWM program. This orientation helped patient-families better understand the program's expectations, and offered an opportunity to evaluate readiness to change, barriers for making lifestyle changes, and mental health problems. This information was used to tailor the intervention to better meet the needs of participating patient-families. When a survey of program characteristics was conducted of the 33 participating sites, this "top-performing site" was the only one to offer such a program orientation session prior to patient-families starting the PWM program. Therefore this program feature was included as part of the "bundle of program enhancements" (BPE) for this proposed pragmatic pilot study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 12 years of age and < 18
* Scheduled for a new patient clinic visit at the multi-component PWM program at CCHMC or HDVCH
* Severe obesity (≥ 120% of the 95th percentile for BMI based on age and gender at time of screening visit)
* Able to understand and complete the consent process
* Have access to a smart phone, device, or computer with a web camera
* Have access to the internet

Exclusion Criteria:

* Lacking capacity to provide informed consent
* Non-English speaking
* Participating in any other weight management program or research study related to weight management
* Have a sibling participating in any other weight management program or research study related to weight management
* Taking anti-obesity medication (Phentermine, Orlistat, Qsymia, Naltrxone-Bupropion, Lorcaserin, others at the discretion of the PI)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One additional participant enrolled to make up for a lost to follow-up.
Period: Overall Study
Arm/Group | Telehealth Intervention | Standard of Care Control
Started | 39 | 22
Completed | 14 | 11
Not Completed | 25 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telehealth Intervention | Standard of Care Control | Total
Number analyzed (Participants) | 39 | 22 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 22 | 61
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.9 [12.5 to 18.0] | 14.8 [12.2 to 17.6] | 14.8 [12.2 to 18.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 28
  Male | 20 | 13 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 35 | 22 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 31 | 16 | 47
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 22 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Implemenmtation of BPE (Bundle of Program Enhancements) in Existing Multi-component PWM Programs
Description: Successful implementation of a "bundle of program enhancements" by existing clinical staff within existing pediatric weight management programs. This success will be defined by ≥80% of randomized intervention group participants and their parent/guardian attending the individual program orientation prior to their initial medical assessment as part of the pediatric weight management program and completing the interactive remote follow-up encounters to achieve the 26 provider contact hours in combination with time spent at clinic visits over the 6 month treatment period.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 39 | 22
Participants | 20 | 12

2. Primary Outcome: Number of Participants Completing Six Month Treatment Period
Description: Completion of the 6 month treatment period will be tracked.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 39 | 22
Participants | 20 | 12

3. Secondary Outcome: Participation Rates in Clinic Visits and Group Sessions
Description: Attendance of participants in each group throughout study period; from baseline visit through 6 month follow up period.
Time Frame: Baseline to 6 months
Population: Number of participants who have baseline data
Measure: Number; unit: participants
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 37 | 21
participants | 37 | 21

4. Secondary Outcome: Change in Percent of the 95th Percentile for Body Mass Index
Description: The health outcome to be evaluated is change in percent of the 95th percentile for body mass index.
Time Frame: 6 months
Population: Intervention of telehealth vs standard of care for change in percent of 95th percentile for body mass index.
Measure: Least Squares Mean (Standard Error); unit: percent of 95th percentile for BMI
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 15 | 10
percent of 95th percentile for BMI | -1.07 (1.90) | -2.35 (2.26)

5. Secondary Outcome: Change in Percentage of Body Fat
Description: The health outcome to be evaluated is change in percent body fat (%).
Time Frame: 6 months
Population: After 6 months of data collection, percent body fat calculations are compared between the two groups
Measure: Median (Inter-Quartile Range); unit: percentage of body fat
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 15 | 8
percentage of body fat | 0.4 [-0.80 to 1.6] | 0.10 [-1.7 to 0.85]

6. Secondary Outcome: Skeletal Muscle Mass Improvement Over Time
Description: The health outcome to be evaluated is change in skeletal muscle mass (kg). An improvement will be indicated by an increase in skeletal muscle mass.
Time Frame: 6 months
Population: Change in skeletal muscle mass after 6 month treatment period in intervention vs control group
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 15 | 8
kg | 0.8 [-0.10 to 2.0] | 0.80 [-0.45 to 1.85]

7. Secondary Outcome: Improvement in Systolic and Diastolic Blood Pressure
Description: The health outcome to be evaluated is change in both systolic and diastolic blood pressure (mmHg).
Time Frame: 6 months
Population: Change in systolic blood pressure and diastolic blood pressure from baseline to 6 month evaluation in intervention participants vs control group participants
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 13 | 6
mmHg
  Systolic Blood Pressure | 2.0 [-3.0 to 8.0] | 2.0 [-8.0 to 8.0]
  Diastolic Blood Pressure | 2.0 [-4.0 to 8.0] | -6.0 [-16.0 to 0.0]

8. Secondary Outcome: Improvement in Lab Values for Serum ALT
Description: The health outcome to be evaluated is the change in the lab value of ALT
Time Frame: 6 months
Population: Change in ALT blood value from baseline to 6 month visit
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 8 | 6
IU/L | 2.00 [-8.0 to 4.5] | 2.00 [-5.0 to 4.0]

9. Secondary Outcome: Change in Triglyceride
Description: Change in triglyceride levels from baseline to 6 months in intervention vs control group participants
Time Frame: 6 months
Population: Change in triglyceride levels from baseline to 6 months in intervention vs control group participants
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 9 | 6
mg/dL | -1.00 [-21.0 to 16.0] | -4.00 [-6.0 to 3.0]

10. Secondary Outcome: Change in Hba1C Levels
Description: Change in Hba1C from baseline to 6 month visit in intervention vs control group
Time Frame: 6 months
Population: Change in Hba1C from baseline to 6 month visit in intervention vs control group
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 8 | 6
percent | -0.05 [-0.15 to 0.15] | 0.15 [0.00 to 0.20]

11. Secondary Outcome: Change in Non-HDL Cholesterol
Description: Change in non-HDL cholesterol from baseline to 6 month visit in intervention vs control group participants
Time Frame: 6 months
Population: Change in non-HDL cholesterol from baseline to 6 month visit in intervention vs control group participants
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 9 | 5
mg/dL | 0.00 [-12.0 to 5.0] | 9.00 [5.0 to 14.0]

12. Secondary Outcome: Change in Fasting Glucose
Description: Change in fasting glucose from baseline to 6 month visit in intervention vs control group participants
Time Frame: 6 months
Population: Change in fasting glucose from baseline to 6 month visit in intervention vs control group participants
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 9 | 6
mg/dL | -3.00 [-4.0 to 1.0] | 7.00 [1.0 to 15.0]

13. Secondary Outcome: Test Whether the Intervention Group Has Greater Rates of Participation and Retention in Standard-of-care Clinic Visits and Group Sessions (if Offered) Compared to the Control Group.
Description: Attendance of participants in each group at 3 month follow up visit
Time Frame: 3 months
Population: Number of participants remaining in study after baseline to 3 month follow up study period
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 27 | 14
Participants | 27 | 14

14. Secondary Outcome: Test Whether the Intervention Group Has Greater Rates of Participation and Retention in Standard-of-care Clinic Visits and Group Sessions (if Offered) Compared to the Control Group.
Description: Attendance of participants in each group at 6 month follow up visit
Time Frame: 6 months
Population: Number of participants remaining at study end point with some amount of data provided
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention | Standard of Care Control
Number analyzed (Participants) | 16 | 12
Participants | 16 | 12

ADVERSE EVENTS:
Time Frame: Each patient was observed for adverse events over their 6 month enrollment period.
Arm/Group | Telehealth Intervention | Standard of Care Control
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/22
Other Adverse Events (participants affected / at risk) | 2/39 | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telehealth Intervention (N=39) | Standard of Care Control (N=22)
Low HDL Cholesterol (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Elevated AST (Blood and lymphatic system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT03939494/Prot_SAP_000.pdf